CLINICAL TRIAL: NCT01741610
Title: Rapid Fluid Administration and the Incidence of Hypotension Induced by Spinal Anaesthesia and Ephedrine Requirement: the Effect of Crystalloid Versus Colloid Coloading
Brief Title: Fluid Coloading and the Incidence of Hypotension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Hakki Unlugenc, Prof Dr., Cukurova University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: HZLTNS97
Record Dates: First submitted 2012-11-15; First posted 2012-12-05 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2014-01

CONDITIONS: Complications; Cesarean Section; Anesthesia; Adverse Effect, Spinal and Epidural; Other Fluid Overload
Keywords: Anaesthesia Spinal; Ephedrine; Fluid Therapy; Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- No coloading (Group E) (Placebo Comparator): Placebo comparator
  Interventions: Biological: Cristalloid and colloid coloading
- Cristalloid (Lactated Ringer) Coloading (Active Comparator): Cristalloid (Lactated Ringer's) Coloading (Group L)
  Interventions: Biological: Cristalloid and colloid coloading
- Colloid (HES) coloading (Active Comparator): Colloid (HES) coloading (Group C)
  Interventions: Biological: Cristalloid and colloid coloading

INTERVENTIONS:
Biological: Cristalloid and colloid coloading — Cristalloid coloading (Group L) Colloid coloading (Group C) No coloading (Group E)Placebo Comparator
  Other Names: Cristalloid coloading (Group L); Colloid coloading (Group C); No coloading (Group E)Placebo Comparator

SUMMARY:
This study was conducted to evaluate the effects of rapid crystalloid (Lactated Ringer's solution) or colloid (hydroxyethyl starch; HES) cohydration with a second intravenous access line on the incidence of hypotension and ephedrine requirement during spinal anaesthesia for caesarean section.

DETAILED DESCRIPTION:
Background: Spinal anaesthesia for caesarean delivery is often associated with hypotension. This study was conducted to evaluate the effects of rapid crystalloid (Lactated Ringer's solution) or colloid (hydroxyethyl starch; HES) cohydration with a second intravenous access line on the incidence of hypotension and ephedrine requirement during spinal anaesthesia for caesarean section.

Methods: We studied 90 women with uncomplicated pregnancies undergoing elective caesarean section under spinal anaesthesia. Intravenous access was established in all with two peripheral intravenous lines, the first being used for the baseline volume infusion. Immediately after induction of spinal anaesthesia, Lactated Ringer's solution (Group L) or HES (Group C) infusions were started at the maximal possible rate via the second line in groups L and C respectively. The third group (Group E) patients received lactated Ringer's solution at a 'keep vein open' rate to maintain the double-blind nature. The incidence of hypotension, ephedrine requirements, total amount of volume and side effects were recorded.

ELIGIBILITY:
Inclusion Criteria:

* elective caesarean section under spinal anaesthesia

Exclusion Criteria:

* Significant coexisting disease such as; pre-eclampsia and hepato-renal disease,
* Pregnancy preinduced hypertension,
* Being in active labour or requiring emergency caesarean section,
* Any contraindication to regional anaesthesia such as local infection or bleeding disorders.

Ages: 19 Years to 46 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2008-10; Primary Completion 2011-08 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Rapid fluid administration and the incidence of hypotension induced by spinal anaesthesia and ephedrine requirement: the effect of crystalloid versus colloid coloading | Four Years
  The primary study endpoint was the ephedrine requirement (incidence of hypotension).

CONTACTS AND LOCATIONS:
Overall Officials: Hakki Unlugenc, Prof Dr, Study Chair — Cukurova University
Locations (1):
- Hakki Unlugenc, Adana, Turkey (Türkiye)

REFERENCES:
- See also: Cukurova University — http://lokman.cukurova.edu.tr